CLINICAL TRIAL: NCT00910468
Title: Robot-Assisted Laparoscopic Myomectomy Is an Improvement Over Laparotomy in Patients With a Limited Number of Fibroids
Status: Completed | Type: Observational
Sponsor: Ascher-Walsh, Charles, M.D. (Individual)
Responsible Party: Char;es Ascher-Walsh, Mount Sinai School of Medicine
Other Study IDs: HSD08-00631
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Fibroid Uterus
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Robot Assisted Laparoscopic Myomectomy
  Interventions: Procedure: Robot-assisted Laparoscopic myomectomy
- Myomectomy via Laparotomy

INTERVENTIONS:
Procedure: Robot-assisted Laparoscopic myomectomy — Robot-assisted Laparoscopic myomectomy
  Groups: Robot Assisted Laparoscopic Myomectomy

SUMMARY:
This is a retrospective, case-control study of 75 patients having undergone a robotic-assisted laparoscopic myomectomy were compared to patients having undergone myomectomy via laparotomy. Both groups had 3 or fewer fibroids confirmed by pre-operative MRI or on final pathology report. Charts were reviewed for surgical and post-operative variables

ELIGIBILITY:
Inclusion Criteria:

* uterus less than or equal to 20 weeks in size by office exam and no greater than three intramural fibroids on pre-operative MRI.

Exclusion Criteria:

* significant medical problems limiting their ability to undergo a prolonged laparoscopic procedure and could not have had previous uterine surgery.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women with fibroid uterus desiring surgical management
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2005-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Post-operative variables, including estimated blood loss, length of stay, days to a regular diet and febrile morbidity | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ascher-Walsh, MD, MPH, Principal Investigator — Mt Sinai School of Medicine, Dept Obstetrics and Gynecology
Locations (1):
- Mount SInai School of Medicine, New York, New York, United States